CLINICAL TRIAL: NCT00581009
Title: The Role of Dopamine Metabolism in the Antidepressant Effects of Sleep Deprivation and Sertraline in Depressed Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joseph Wu, Professor of Psychiatry & Human Behavior, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20011616
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Sleep deprivation; antidepressant; depression; chronobiological
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Sleep Deprivation; Depression | interventions — Sertraline; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Chronobiological augmentation (Experimental): chronobiological augmentation group
  Interventions: Other: chronobiological augmentation
- Medication only (Experimental): medication only group
  Interventions: Drug: sertraline, lithium
- MDD Mechanism (Experimental)
  Interventions: Radiation: one night of sleep deprivation and two FDG PET scans

INTERVENTIONS:
Other: chronobiological augmentation — Sleep deprivation for one night, Chronobiological augmentation consists of partial sleep phase advance for three nights and Light therapy for two hours for three days
  Arms: Chronobiological augmentation
Drug: sertraline, lithium — Antidepressant, Subjects will be started on a serotonin specific reuptake inhibitor (SSRI), sertraline 100 mg (50mg hs x 2) daily or other SSRI's such as Paxil 20 mg or Prozac 20 mg daily and continue treatment for seven weeks.
  Mood stabilizer, subjects will be treated with lithium 450 mg twice a day or another mood stabilizer such as depakote or valproate and continue treatment for seven weeks.
  Other Names: Zoloft; Lithium
  Arms: Medication only
Radiation: one night of sleep deprivation and two FDG PET scans — MDD Mechanism Only depressed subjects will have two FDG PET scans consisting of a baseline FDG PET scan and a sleep deprived FDG PET scan. One night of regular sleep,one night of sleep deprivation and one night of recovery sleep for a total of four nights at a sleep laboratory facility.
  Arms: MDD Mechanism

SUMMARY:
This study evaluates the efficacy of sleep deprivation treatment in accelerating antidepressant responses when administered during the first week of medications and augmenting a sustained response with chronobiological interventions. Sleep deprivation and chronobiological augmentation may offer a rapid and sustained antidepressant response in mood disorder patients treated with medication, sleep deprivation, bright light therapy and sleep phase advance compared with medication only. The chronobiological treatment is rapid, non-invasive and has few side effects and could be of significant clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include:

1. Subjects must be English speaking
2. Subjects must have either bipolar or unipolar depression diagnosis or be a normal control.
3. Subjects must be between : 18 to 75

Non-English speaking subjects will be excluded since scales for measuring depression have not been validated in languages other than English.

Exclusion Criteria:

Exclusion criteria include:

1. Suicidality, or psychosis
2. Unstable medical conditions
3. Epilepsy, serious head injury, or other significant neurological disorders
4. Dementia, mental retardation (moderate or severe), coma
5. Prior exposure to radiation which might cause the subject to exceed standard guidelines
6. Substance abuse or alcoholism in the past six months
7. Unreliability or inability to adhere to the requirements of the study
8. Irregular sleep-wake schedules (nightshift, jet lag)
9. Use of CNS medications which may affect sleep or functional brain imaging (i.e., use of sleeping pills, antidepressants or other mood stabilizers or other medications which may affect the sleep EEG)
10. Sleep apnea, periodic limb movements of sleep, narcolepsy, circadian sleep phase disorders
11. Donation or loss of blood (>400 ml) within the past month
12. Current or very recent intercurrent illnesses, painful conditions or other disorders, which in the judgement of the investigators, might invalidate the scientific goals of the study or pose undesirable difficulties or risks for the subject.
13. Hamilton Rating Scale of Depression (HRSD-17 items)<17 unless subject is a normal control subject.
14. Pregnancy or breast feeding
15. Individuals who would be unable to undergo a magnetic resonance imaging (MRI) scan, for example, individuals who suffer from claustrophobia, or who have metal clips in their body.
16. Unable to cease taking psychoactive medications which are not part of this protocol (2-5 weeks) prior to PET scans.
17. Patients with previous history of significant adverse reactions to sertraline or sertraline-like drugs or other SSRI's such as Paxil or Prozac
18. Subjects with diagnosis of eating disorder/bulimia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2001-05-30 (Actual); Primary Completion 2011-12-09 (Actual); Study Completion 2011-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry F Chaitin, M.D., Study Chair — University of California, Irvine
Locations (2):
- United States (2):
  - University of California, Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication Only Group: medication only group
  Medication as usual, which included sertraline, lithium: Antidepressant, Subjects will be started on a serotonin specific reuptake inhibitor (SSRI), sertraline 100 mg (50mg hs x 2) daily or other SSRI's such as Paxil 20 mg or Prozac 20 mg daily and continue treatment for seven weeks.
  Mood stabilizer, subjects will be treated with lithium 450 mg twice a day or another mood stabilizer such as depakote or valproate and continue treatment for seven weeks.
- Chronobiological Augmentation Group: chronobiological augmentation group
  Chronobiological augmentation consists of sleep deprivation for one night, partial sleep phase advance for three nights, and light therapy for two hours for three days
Period: Overall Study
Arm/Group | Medication Only Group | Chronobiological Augmentation Group
Started | 17 | 32
Sample Recruitment | 17 | 32
Completed | 17 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All bipolar depressed subjects
Groups:
- Chronobiological Augmentation: chronobiological augmentation group
  chronobiological augmentation: Chronobiological augmentation consists of sleep deprivation for one night, partial sleep phase advance for three nights and ight therapy for two hours for three days
- Medication Only: medication only group
  medication as usual, including: sertraline, lithium: Antidepressant, Subjects will be started on a serotonin specific reuptake inhibitor (SSRI), sertraline 100 mg (50mg hs x 2) daily or other SSRI's such as Paxil 20 mg or Prozac 20 mg daily and continue treatment for seven weeks.
  Mood stabilizer, subjects will be treated with lithium 450 mg twice a day or another mood stabilizer such as depakote or valproate and continue treatment for seven weeks.
- Total: Total of all reporting groups
Arm/Group | Chronobiological Augmentation | Medication Only | Total
Number analyzed (Participants) | 32 | 17 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 17 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13) | 40 (14) | 39.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 22 | 7 | 29
Region of Enrollment [Number; unit: participants]
  United States | 32 | 17 | 49

OUTCOME MEASURES:

1. Primary Outcome: Total Score on the Hamilton Rating Score for Depression (HRSD) - 21 Item Version
Description: Difference in HRSD between the chronobiological augmentation therapy and medication only groups across the first 7 days, and up to 7 weeks of treatment. The 21-item HRSD has a range of 0 to 66, with a higher score indicating more severe depression.
Time Frame: within the first seven days up to 7 weeks (plus or minus 1 day) after sleep deprivation and chronobiological therapy
Population: Bipolar disorder subjects
Measure: Mean (Standard Deviation); unit: Total score on a scale
Groups:
- Medication Only: medication only group
  sertraline, lithium: Antidepressant, Subjects will be started on a serotonin specific reuptake inhibitor (SSRI), sertraline 100 mg (50mg hs x 2) daily or other SSRI's such as Paxil 20 mg or Prozac 20 mg daily and continue treatment for seven weeks.
  Mood stabilizer, subjects will be treated with lithium 450 mg twice a day or another mood stabilizer such as depakote or valproate and continue treatment for seven weeks.
Arm/Group | Chronobiological Augmentation | Medication Only
Number analyzed (Participants) | 32 | 17
Total score on a scale
  Baseline | 19 (6.7) | 18.5 (7.1)
  Day 7 | 10.2 (7.3) | 14.4 (8)
  Week 7 | 10.1 (9.6) | 15.2 (10.2)
Statistical Analysis 1: Comparison: Chronobiological Augmentation vs Medication Only; Test type: Equivalence — repeated measure ANOVA; p < 0.05, ANOVA; t-value = 3.34

ADVERSE EVENTS:
Arm/Group | Chronobiological Augmentation | Medication Only
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/17
Other Adverse Events (participants affected / at risk) | 2/32 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronobiological Augmentation (N=32) | Medication Only (N=17)
brief hypomanic switch (Psychiatric disorders) | 2 (2) | 0 (0) — brief hypomanic period including pressured speech and elevated mood

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No